CLINICAL TRIAL: NCT00926653
Title: Anterior Cingulate Activation in Geriatric Depression
Brief Title: Assessing Anterior Cingulate Brain Activity in People With Late-Life Depression
Status: Completed | Type: Observational
Sponsor: Weill Medical College of Cornell University (Other)
Responsible Party: Sponsor
Other Study IDs: K23MH074818 (NIH); DATR AK-TNGP1
Record Dates: First submitted 2009-06-22; First posted 2009-06-23 (Estimated); Last update posted 2015-08-11 (Estimated); Status verified 2015-08

CONDITIONS: Depression
Keywords: Geriatric Depression
MeSH Terms: conditions — Depression | interventions — Escitalopram

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Depressed: Elderly participants with depression
  Interventions: Drug: Escitalopram
- Control: Elderly participants who have never experienced depression

INTERVENTIONS:
Drug: Escitalopram — 10 to 20 mg daily as part of another study in which participants are enrolled
  Other Names: Lexapro
  Groups: Depressed

SUMMARY:
This study will examine differences in activity of the anterior cingulate cortex, a brain area involved in emotion and cognitive regulation, between older adults with and without depression.

DETAILED DESCRIPTION:
Older adults with depression often also suffer from executive dysfunction-problems with planning, impulse control, and reasoning. Executive dysfunction in older adults predicts poor or delayed response to antidepressant treatment and has been associated with early relapse and recurrence of late-life major depression. Functional magnetic resonance imaging (fMRI) is a scan that can measure the activity of someone's brain while that person performs tasks. So far, no fMRI studies investigating cerebral activation patterns in late-life depression have been published. In this study, people will undergo fMRI while they are performing an executive function task. Older adults with late-life depression and older adults without depression will be tested and compared in order to identify the areas and patterns of brain activity underlying executive dysfunction in late-life depression.

Participation in this study will consist of one study visit, during which participants will undergo an fMRI scan that will last 60 to 90 minutes. While being scanned, participants will perform cognitive tasks that involve pressing buttons in response to words viewed on a screen.

ELIGIBILITY:
Inclusion Criteria for Depressed Participants:

* Diagnosis of major depression by DSM-IV criteria
* Mini-Mental State Examination (MMSE) score greater than 24
* Severity score of 17 or higher on the 21-item Hamilton Depression Rating Scale score (HDRS) during the index episode
* Residence less than a 45-minute drive from New York Hospital-Westchester Division

Exclusion Criteria for Depressed Participants:

* Presence of psychotic depression, as defined by Research Diagnostic Criteria and DSM-IV
* History of psychiatric disorders other than unipolar major depression (people with bipolar disorder and dysthymia will be excluded)
* Presence of dementing disorders
* Acute or severe medical illness, such as the following: delirium; metastatic cancer; decompensated cardiac, liver, or kidney failure; major surgery; or cerebrovascular accident or myocardial infarction 3 months prior to study entry
* Receiving drugs known to cause depression, including reserpine, alpha-methyl-dopa, and steroids
* Requires concomitant treatment with other psychotropics, including antipsychotic medications, lithium salts, stimulants, valproic acid, carbamazepine, or gabapentin
* Severe aphasia interfering with communication
* Contraindications to magnetic resonance (MR) scanning, such as implanted metal, claustrophobia, or weight greater than or equal to 300 lbs

Inclusion Criteria for Age-Matched Non-Psychiatric Comparison Sample:

* MMSE score greater than 24

Exclusion Criteria for Age-Matched Non-Psychiatric Comparison Sample:

* History of psychiatric disorder
* Presence of dementing disorders
* Acute or severe medical illness, such as the following: delirium; metastatic cancer; decompensated cardiac, liver, or kidney failure; major surgery; or cerebrovascular accident or myocardial infarction 3 months prior to study entry
* Receiving drugs known to cause depression, including reserpine, alpha-methyl-dopa, and steroids
* Current treatment with psychotropics
* Severe aphasia interfering with communication
* Contraindications to MR scanning, such as implanted metal, claustrophobia, or weight greater than or equal to 300 lbs

Ages: 60 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Depressed and control participants are recruited from the community, with additional depressed participants recruited from a geriatric outpatient clinic at New York Presbyterian/Weill Cornell Medical College.
Sampling Method: Non-Probability Sample
Enrollment: 76 (Actual)
Dates: Start 2005-07; Primary Completion 2010-05 (Actual); Study Completion 2010-05 (Actual)

PRIMARY OUTCOMES:
Cerebral activation, as measured using functional magnetic resonance imaging (fMRI) | Average of a 2 hour MRI session

CONTACTS AND LOCATIONS:
Overall Officials: Faith M. Gunning-Dixon, PhD, Principal Investigator — Weill Medical College of Cornell University
Locations (1):
- New York Presbyterian-Weill Cornell Medical College, White Plains, New York, United States